CLINICAL TRIAL: NCT05499585
Title: Treating Pediatric NAFLD with Nutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jeffrey B. Schwimmer, MD, Principal Investigator, Professor of Clinical Pediatrics, University of California, San Diego
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 803602
Record Dates: First submitted 2022-08-10; First posted 2022-08-12 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Liver Diseases; Liver Fat; Hepatic Steatosis; Nutritional and Metabolic Disease
Keywords: child; adolescent; nutrition; liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Liver Diseases; Fatty Liver; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm One (Other): Habitual diet for 12 weeks followed by experimental diet for 12 weeks
  Interventions: Other: Whole Dairy

INTERVENTIONS:
Other: Whole Dairy — 2 1/2 servings of whole dairy per day

SUMMARY:
This is a proof of concept clinical trial to compare daily intake of at least 20 grams of whole dairy fat vs habitual diet on hepatic steatosis in children with NAFLD.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is the most common chronic liver disease in children, estimated to be present in 5-10% of all children in the United States. NAFLD is a growing cause of cirrhosis and liver cancer. There is not yet an FDA approved treatment for NAFLD. Guidelines recommend improvement in diet at the first line of treatment; however, there is no consensus as to what that diet should be. General health guidelines recommend nonfat or low fat dairy over whole dairy after age 2. Limited studies have suggested that whole dairy may be better for people with NAFLD.

This study will test the effect of whole dairy on liver fat in children age 10-17 with NAFLD. As a baseline, the investigators will measure liver fat (using MRI) at 2 time points separated by 12 weeks to establish the current amount of liver fat. The children will be instructed to incorporate 2 ½ servings of whole dairy (as milk and/or yogurt provided by the study will provide) into their daily diet. After 12 weeks, the investigators will measure liver fat with MR and labs to assess safety and further evaluate the liver.

ELIGIBILITY:
Inclusion Criteria:

* Age 10 through 17 years
* NAFLD
* ALT of ≥ 40 U/L
* MRI-PDFF ≥ 8%
* Ability and willingness of legal guardian and participant to provide written, informed consent

Exclusion Criteria:

Competing Health Conditions

* Participants with a history of health issues that make it unsafe for them to participate in the opinion of the investigator
* Type 1 or Type 2 Diabetes
* LDL-cholesterol > 160 mg/dL
* Evidence of other chronic liver disease (alcohol liver disease, alcohol related liver disease, hepatitis C, chronic hepatotoxic drug use, mitochondrial diseases, autoimmune liver disease, wilson's disease)
* History of bariatric surgery or planning to undergo bariatric surgery during the study duration
* Participant with a history of conditions affecting digestion and/or absorption

Intervention

* Inability or refusal to consume dairy
* Cow's milk protein allergy
* Lactose intolerance

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Change in hepatic steatosis measured by liver MRI-PDFF | Baseline to 12 weeks and 12 weeks to 24 weeks
  The primary outcome for the 24 week study is to compare daily intake of at least 20 grams of whole dairy fat vs habitual diet on hepatic steatosis in children with NAFLD

SECONDARY OUTCOMES:
Change in serum alanine transaminase (ALT) | Baseline, week 12 and week 24
  ALT will be measured and compared
Change in serum aspartate transaminase (AST) | Baseline, week 12 and week 24
  AST will be measured and compared
Change in serum gamma-glutamyl transpeptidase (GGT) | Baseline, week 12 and week 24
  GGT will be measured and compared
Change in serum total cholesterol | Baseline, week 12 and week 24
  Serum total cholesterol will be measured and compared
Change in serum LDL-cholesterol | Baseline, week 12 and week 24
  Serum LDL-cholesterol will be measured and compared
Change in serum HDL-cholesterol | Baseline, week 12 and week 24
  Serum HDL-cholesterol will be measured and compared
Change in serum triglycerides | Baseline, week 12 and week 24
  Serum triglycerides will be measured and compared
Change in plasma fatty acid levels | Baseline, week 12 and week 24
  Plasma fatty acid levels will be measured and compared
Change in subcutaneous adipose tissue (SCAT) | Baseline, week 12 and week 24
  SCAT will be measured and compared
Change in visceral adipose tissue (VAT) | Baseline, week 12 and week 24
  VAT will be measured and compared

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Schwimmer, MD, Principal Investigator — UC San Diego
Locations (1):
- UC San Diego, La Jolla, California, United States